CLINICAL TRIAL: NCT04270825
Title: Group Treatment for Hoarding Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Brittany Mathes, Graduate Student, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018.26389
Record Dates: First submitted 2019-03-25; First posted 2020-02-17 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Hoarding Disorder
MeSH Terms: conditions — Hoarding Disorder | interventions — adenylate isopentenyltransferase

STUDY DESIGN:
Intervention Model Description: Participants will receive a novel treatment for hoarding disorder.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT with IPT (Experimental): Group CBT with IPT will consist of 20 weekly two-hour sessions and has been developed for the proposed study based on the protocols for group CBT for HD and group IPT. Treatment includes strategies from CBT, including cognitive restructuring, behavioral exposures, and organizational strategies, as well as strategies from IPT, including role-play, interpersonal skills building, communication analysis, and decision analysis.
  Interventions: Behavioral: Group CBT with IPT

INTERVENTIONS:
Behavioral: Group CBT with IPT — Group treatment designed to target relationships with both possessions and people.

SUMMARY:
This study assesses the effectiveness of a novel group treatment for hoarding disorder.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate the effectiveness of a novel group treatment for hoarding disorder. Participants will be randomized to receive either treatment as usual (cognitive behavioral therapy: CBT) or treatment as usual augmented by interpersonal psychotherapy (IPT). It is hypothesized that group CBT with IPT will result in greater decreases in hoarding symptoms, as compared to standard group CBT. It is further hypothesized that CBT with IPT will result in greater reductions in object attachment and maladaptive beliefs about relationships with others, as well as greater increases in interpersonal attachment.

ELIGIBILITY:
Inclusion Criteria:

-Clinical diagnosis of HD

Exclusion Criteria:

* Evidence of a severe mental illness or substance use disorder that would impede the completion of the treatment
* Current receipt of CBT for HD
* Initiation of new psychotropic medications for symptoms of HD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in Hoarding Rating Scale (HRS) | Baseline, 10 weeks, 20 weeks, 24 weeks
  The Hoarding Rating Scale is a commonly used measure of hoarding symptoms in which participants rate the severity of their symptoms. Minimum score is 0 and maximum score is 40. Higher scores indicate more severe/worse symptoms.
Changes in Reciprocal Attachment Questionnaire Adapted (RAQ-A) | Baseline, 10 weeks, 20 weeks, 24 weeks
  The Reciprocal Attachment Questionnaire Adapted assesses attachment to one's belongings, with higher scores indicating greater attachment to possessions (i.e., worse outcome). Minimum score is 75 and maximum score is 375.
Changes in Adult Attachment Scale (AAS) | Baseline, 10 weeks, 20 weeks, 24 weeks
  The AAS is a measure of two dimensions proposed to underlie interpersonal attachment security: anxiety and avoidance. Higher scores indicate worse outcomes. Minimum score is 0 and maximum score is 72.
Changes in Interpersonal Needs Questionnaire (INQ) | Baseline, 10 weeks, 20 weeks, 24 weeks
  The INQ is a measure of two interpersonal risk factors, namely perceived burdensomeness and thwarted belongingness, with higher scores indicating higher levels of each construct (i.e., worse outcome). Minimum score is 15 and maximum score is 105.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared.